CLINICAL TRIAL: NCT01956019
Title: Feasibility Study to Compare Early Response Assessment and Planning Volumes With Contrast-enhanced Computed Tomography (CT), MRI Including Diffusion Weighted MRI (DWI) and Dynamic-contrast Enhanced (DCE) MRI in Patients With Limb Sarcoma Undergoing Pre-operative Radiotherapy
Brief Title: MRI in Pre-operative Radiotherapy for Soft Tissue Sarcoma: MISTS Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Emmie Taylor, Clinical Trials Project Manager, The Christie NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10_RADIO_96
Record Dates: First submitted 2013-04-26; First posted 2013-10-08 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI scanning (Experimental): patients undergo special MRI techniques (DWI-MRI and DCE-MRI) after their routine MRI examinations while undergoing routine radiotherapy. 3 lots of scans in total. They will also have a blood test.
  Interventions: Device: MRI scanning

INTERVENTIONS:
Device: MRI scanning

SUMMARY:
This study will use diffusion weighted MRI (DWI MRI) and dynamic-contrast enhanced MRI (DCE MRI) techniques to detect changes in sarcoma tumour vasculature. The main aims of this study are to correlate histological response of soft tissue sarcoma after pre-operative radiotherapy with several pre-treatment DCE and DWI MRI parameters and to assess the impact of these on early response prediction. Detected changes may reflect the sensitivity of the tumour to radiotherapy and may be associated with long term outcomes after treatment.

15 patients normally having pre-operative radiotherapy as part of their sarcoma treatment will be recruited to this study.

Patients will have an additional three specialised MRI scans: one prior to the start of radiotherapy, one during the second week of radiotherapy while on treatment and one scan a week before surgery but after the completion of radiotherapy.

Post-operatively, results of the histological examination of the sarcoma will be correlated to both the MRI scan data and outcomes after treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of intermediate/high grade soft tissue sarcoma (STS)
* Patients must be suitable for treatment with preoperative radiotherapy and radical surgery
* Standard radiological assessments (CT or MRI) may have already been performed but must be done within 4 weeks of starting radiotherapy
* Patient must have measurable disease on CT/MRI imaging
* ECOG performance status 0-2
* Adequate pre-treatment haematological and biochemical parameters
* Age greater than or equal to 18 years
* No significant co-morbidity thereby excluding patient from having radical treatment.
* No previous treatment for diagnosis of STS including neo-adjuvant chemotherapy
* Women of child bearing age MUST have a negative pregnancy test prior to study entry and be using an adequate contraception method unless child bearing potential has been terminated by surgery/radical radiotherapy
* Patients must have given written informed consent

Exclusion Criteria:

* Patients with cardiac pacemakers, cochlear implants, intraocular foreign bodies or any other MRI incompatibility factors (e.g. recent surgery).
* Patients with a known history of anaphylactic reaction to contrast material for MRI
* Previous administration of gadoxetic acid or other contrast material 24hr prior to or after the MRI
* Any evidence of severe or uncontrolled systemic diseases which, in the view of the investigator, makes it undesirable for the patient to participate in the trial
* Evidence of significant clinical disorder or laboratory finding which, in the opinion of the investigator makes it undesirable for the patient to participate in the trial
* Any other serious uncontrolled medical conditions
* Clinical evidence of metastatic disease
* Any pregnant or lactating woman
* Any patient with a medical or psychiatric condition that impairs their ability to give informed consent
* Evidence of impaired renal function, serum creatinine >1.5x upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Correlate histological response of soft tissue sarcoma after pre-operative radiotherapy with pre-treatment DWI and DCE-MRI parameters. | average of 9 weeks including radiotherapy up to one week before surgery
  The hypothesis is that quantitative biomarkers from DWI and DCE MRI can not only be produced with high spatial resolution in soft tissue sarcoma, but that these imaging biomarkers will correlate with histological and histochemical features of the tumour and will provide information to support the prediction of regional response to radiotherapy.

SECONDARY OUTCOMES:
early response prediction of treatment using functional parameters of in-treatment imaging with DWI and DCE-MRI (e.g. relative change in apparent diffusion coefficient values) | following surgery at week 7
accuracy of outlining treatment volumes using STIR. T1W, T2W and DWI MRI compared to standard planning CT and loco-regional control patterns | 3 month follow up visit
local recurrence patterns with pre-treatment functional MRI. | 3 timepoints for scans over 6 weeks of treatment
  Within our study, these patients would have an additional three specialised MRI scans: one prior to the start of radiotherapy, one during the second week of radiotherapy while on treatment and one scan the week before the operation after the completion of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Manoharan, Study Chair — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom